CLINICAL TRIAL: NCT00658346
Title: Molecular Diversity of HIV-1 Group O Strains and Treatment Management in Cameroon
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 12168 DYNA M-O
Record Dates: First submitted 2008-04-11; First posted 2008-04-15 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: HIV Infections
Keywords: HIV-1 group O; HIV-1 group M; Cameroon; HIV-1 infection; treatment naïve
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma and mononucleus cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: HIV-1 group O infected patients
  Interventions: Drug: Treatment initiation for HIV-1 group O infected patients
- 2: HIV-1 group M infected patients
  Interventions: Drug: Treatment initiation for HIV-1 group M infected patients

INTERVENTIONS:
Drug: Treatment initiation for HIV-1 group O infected patients — The first line regimen is adapted according to the hemoglobin level and the AgHBs status :
  * If Hb > 8 g/ml and negative AgHBs : AZT-3TC (DUOVIR) + LPV/RTV (ALUVIA)
  * If Hb <= 8 g/ml and negative AgHBs : TDF-3TC (LAMIVIR-S) + LPV/RTV (ALUVIA)
  * If positive AgHBs : TDF + 3TC + LPV/RTV (ALUVIA)
  Groups: 1
Drug: Treatment initiation for HIV-1 group M infected patients — The first line regimen is adapted according to the hemoglobin level and the AgHBs status :
  * If Hb > 8 g/ml and negative AgHBs : AZT-3TC (DUOVIR) + LPV/RTV (ALUVIA)
  * If Hb <= 8 g/ml and negative AgHBs : TDF-3TC (LAMIVIR-S) + LPV/RTV (ALUVIA)
  * If positive AgHBs : TDF + 3TC + LPV/RTV (ALUVIA)
  Groups: 2

SUMMARY:
Infections with HIV-1 group O are found in 1 to 3 % of persons living with HIV in Cameroon. The natural history and treatment response is not well understood. The natural resistance to non nucleoside reverse transcriptase inhibitors and their possible low sensitivity to protease inhibitors complicate the choice of an adequate treatment options.

This observational study is aimed at evaluating the antiretroviral treatment response of HIV-1 group O infected patients in comparison with HIV-1 group M infected patients. The proposed standardized follow-up will facilitate a better understanding of the natural history and treatment specificities to improve the patients management.

This is a non randomized study, open label, with standardized follow-up. A total of 171 patients

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 group O or group M infection
* No history of antiretroviral treatment (except for PMTCT)
* Criteria for treatment initiation according to the Cameroons national guidelines

Exclusion Criteria:

* Ongoing traditional treatment which could interfere with hepatic function
* Ongoing treatment with rifabutin, rifampicin or rifampin
* Acute hepatitis B infection
* Pregnancy or lactating mother
* HIV-1 group O and group M co-infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1 infected patients coming for medical care in four treatment centers in Yaounde.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2010-06; Primary Completion 2015-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with plasmatic HIV viral load bellow 60 copies / ml | 48 weeks

SECONDARY OUTCOMES:
Proportion of patients with plasmatic HIV viral load bellow 60 copies / ml | 24 and 96 weeks
Early and late slope of viral load decrease | between weeks 2 and 12, and week 24
Early and late slope of CD4 counts increase | between weeks 2 and 12, and week 24
Proportion of patients with a stabilized CD4 counts gain over 50% | 96 weeks
Time to virological failure | Through out the trial
Resistance mutation profile when virological failure | Through out the trial
Clinical evaluation : proportion of adverse events, AIDS related events, deaths, morphologic modification | Through out the trial

CONTACTS AND LOCATIONS:
Locations (2):
- Cameroon (2):
  - Hôpital Central, Yaoundé
  - Hôpital de la CNPS, Yaoundé

REFERENCES:
- [Derived] Kouanfack C, Unal G, Schaeffer L, Kfutwah A, Aghokeng A, Mougnutou R, Tchemgui-Noumsi N, Alessandri-Gradt E, Delaporte E, Simon F, Vray M, Plantier JC; ANRS 12168 DynaMO Study. Comparative Immunovirological and Clinical Responses to Antiretroviral Therapy Between HIV-1 Group O and HIV-1 Group M Infected Patients. Clin Infect Dis. 2020 Mar 17;70(7):1471-1477. doi: 10.1093/cid/ciz371. PMID 31063537